CLINICAL TRIAL: NCT06708247
Title: Peri-implant Reconstructive Therapy with Tuberosity Bone with and Without Electrolytic Cleaning in the Surgical Management of Peri-implantitis: a Randomized Clinical Trial.
Brief Title: Reconstructive Therapy for Peri-implantitis Using Tuberosity Bone with or Without Electrolytic Cleaning: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilniaus Implantologijos Centro (VIC) Klinika (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUBER-GALVO-RCT
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Peri-implantitis; Peri-Implant Health; Peri-Implantational Loss; Peri-Implantation Loss
Keywords: peri-implantits; dental implants; bone grafting; Electrolytic cleaning
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: This study follows a parallel interventional model where participants are randomly assigned to one of two groups. The control group receives standard peri-implant reconstructive therapy involving mechanical debridement and bone grafting with autogenous tuberosity bone. The test group undergoes the same reconstructive therapy but includes an additional intervention of electrolytic cleaning for implant surface decontamination. Both groups are monitored concurrently over a 12-month period to assess clinical and radiographic outcomes, such as probing pocket depth reduction and bone regeneration. This model allows for a direct comparison of treatment efficacy between the two intervention strategies.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Peri-implant Reconstructive Therapy (Active Comparator): Participants in this arm receive standard peri-implant reconstructive therapy for the management of peri-implantitis. This includes mechanical debridement of the implant surface, bone grafting using autogenous bone from the tuberosity, and the use of a resorbable collagen membrane to promote bone regeneration. The intervention aims to reduce inflammation, improve bone regeneration, and stabilize the implant site.
  Interventions: Procedure: Standard Peri-implant Reconstructive Surgery
- Peri-implant Reconstructive Therapy with Electrolytic Cleaning (Experimental): Participants in this arm undergo peri-implant reconstructive therapy combined with electrolytic cleaning for enhanced decontamination of the implant surface. This includes mechanical debridement, electrolytic cleaning to remove biofilm and contaminants while preserving the implant surface, followed by bone grafting using autogenous bone from the tuberosity and coverage with a resorbable collagen membrane. This intervention is intended to improve clinical outcomes, enhance bone regeneration, and achieve better implant stability compared to the standard therapy alone.
  Interventions: Procedure: Electrolytic Cleaning with Peri-implant Reconstructive Surgery

INTERVENTIONS:
Procedure: Standard Peri-implant Reconstructive Surgery — This intervention involves standard peri-implant reconstructive surgery without the additional step of electrolytic cleaning. The procedure includes mechanical debridement of the implant surface to remove biofilm, followed by bone grafting using autogenous bone harvested from the tuberosity and coverage with a resorbable collagen membrane for bone regeneration and stabilization of the implant.
  Arms: Standard Peri-implant Reconstructive Therapy
Procedure: Electrolytic Cleaning with Peri-implant Reconstructive Surgery — This intervention involves peri-implant reconstructive surgery with an added step of electrolytic cleaning for enhanced implant surface decontamination. The procedure starts with mechanical debridement of the implant surface, followed by the use of an electrolytic cleaning device to remove biofilm and contaminants without damaging the implant surface. This is then followed by bone grafting using autogenous tuberosity bone and coverage with a resorbable collagen membrane to promote bone regeneration and implant stability.
  Arms: Peri-implant Reconstructive Therapy with Electrolytic Cleaning

SUMMARY:
This study aims to evaluate the effectiveness of two surgical approaches for managing peri-implantitis, a condition characterized by inflammation and bone loss around dental implants. Participants will be randomly assigned to one of two groups: one group will receive standard peri-implant reconstructive therapy using bone grafts from the tuberosity region, and the other group will undergo the same treatment with the addition of electrolytic cleaning to decontaminate the implant surface. The primary objective is to determine whether adding electrolytic cleaning improves treatment outcomes by promoting better decontamination and bone regeneration. Clinical assessments, including probing depth measurements and radiographic analysis, will be performed at baseline and at follow-up intervals over 12 months. The study's hypothesis is that the use of electrolytic cleaning alongside standard reconstructive therapy will result in superior clinical and radiographic outcomes compared to the standard method alone.

DETAILED DESCRIPTION:
This randomized clinical trial investigates the effectiveness of reconstructive therapy for peri-implantitis using autogenous bone grafts from the tuberosity, with and without the addition of electrolytic cleaning for implant surface decontamination. Peri-implantitis, an inflammatory condition that results in bone loss around dental implants, poses significant challenges for successful long-term management. Traditional treatment methods focus on mechanical decontamination and bone regeneration, but the outcomes have been inconsistent due to difficulties in achieving thorough surface cleaning without damaging the implant.

This study involves patients diagnosed with peri-implantitis who will be randomly assigned to either the control group or the test group. The control group will undergo conventional treatment, which includes mechanical debridement and grafting with autogenous bone harvested from the tuberosity, covered by a resorbable collagen membrane. The test group will receive an additional step of electrolytic cleaning using a novel electrochemical device designed to decontaminate the implant surface without causing structural damage. This method leverages reactive oxygen species to aid in biofilm disruption and removal.

The trial's primary outcome measures include the reduction in probing pocket depth (PPD) and bleeding on probing (BOP) as well as radiographic assessments of bone regeneration at various time points, up to 12 months post-surgery. Secondary outcomes include patient-reported pain levels, surgical site healing, and the overall stability of bone and soft tissue.

Pre-surgical procedures involve thorough oral hygiene protocols, mechanical debridement, and local application of chlorhexidine and antibiotics. Surgical treatment follows standard implant exposure and flap design techniques, with bone grafts obtained from the tuberosity. For the test group, electrolytic cleaning will be performed prior to graft placement. Post-surgical care includes antibiotics, pain management, and specific oral hygiene instructions to ensure optimal healing.

The study seeks to address the hypothesis that incorporating electrolytic cleaning enhances implant surface decontamination, thus improving clinical outcomes and facilitating more predictable bone regeneration. The findings aim to contribute to the growing body of literature on peri-implantitis management and provide evidence for more effective treatment strategies that preserve implant integrity and support long-term success.

ELIGIBILITY:
Inclusion Criteria:

Participants aged 18 years or older.

Diagnosed with peri-implantitis, characterized by:

Bleeding on probing (BOP) around dental implants. Probing pocket depths (PPD) greater than 6 mm. Implants in function for over 1 year with progressive bone loss exceeding 3 mm. Initial screening confirmed by panoramic radiographs, cone-beam computed tomography (CBCT), and clinical diagnosis.

_____________________________________________

Exclusion Criteria:

Individuals with uncontrolled medical conditions or systemic diseases. Pregnant women. Smokers who smoke more than 10 cigarettes per day. Presence of implant mobility. Situations where the removal of the implant suprastructure is not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) | 12 months
  The primary outcome measure for this study is the reduction in probing pocket depth (PPD) at a 12-month follow-up. PPD is measured at four sites (mesial, distal, buccal, and lingual) around the affected implants to assess the success of treatment in reducing the depth of periodontal pockets. A significant decrease in PPD indicates effective treatment and improved implant health. Clinical probing is performed by a blinded examiner using a standardized periodontal probe to ensure consistency and reliability. Measurements taken at baseline and at 12 months post-surgery will be compared to evaluate the effectiveness of both the standard reconstructive therapy and the therapy with added electrolytic cleaning.

SECONDARY OUTCOMES:
Bone Regeneration Assessed via Radiographic Analysis | 12 months
  Bone regeneration is assessed using standardized radiographic analysis to measure changes in bone levels around the treated implants. Radiographs taken at baseline and at the 12-month follow-up will be analyzed to quantify the amount of new bone formed. Measurements will be conducted at four points (mesial, distal, buccal, and lingual) relative to the implant shoulder. This outcome helps determine the efficacy of the interventions in supporting bone regeneration and stabilizing the implant environment.
Bleeding on Probing (BOP) | 12 months
  This outcome measures the presence of bleeding on probing around the treated implants at baseline and 12 months post-surgery. BOP is a key indicator of gingival inflammation and peri-implant health. Reduction in BOP signifies improved periodontal status and successful treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- VIC Clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) related to primary and secondary outcome measures, including clinical measurements, radiographic analysis results, and probing depths. Data will be made available upon reasonable request and approval by the corresponding author for research purposes.
Supporting Information: Study Protocol
Time Frame: Data will be available starting 6 months after publication of the main study results. Data will be available for a period of 5 years after the initial release.
Access Criteria: Qualified researchers with a valid research proposal related will be able to access the de-identified individual participant data (IPD) and supporting information. Researchers must submit a written request to the corresponding author, detailing the purpose and methodology of their proposed study. Access will be granted upon approval by the research team and will require a signed data use agreement to ensure confidentiality and proper data usage. Data will be provided in a secure format through an encrypted electronic transfer or a secure data-sharing platform.